CLINICAL TRIAL: NCT04333433
Title: A Prospective, Concurrent Controlled, Open-Label, Multicenter Clinical Study to Assess the Long-Term Safety of the PRESERFLO® MicroShunt in Subjects With Primary Open-Angle Glaucoma Who Have Completed Participation in the INN-005 Randomized Controlled Study.
Brief Title: PRESERFLO® MicroShunt Extension Study
Status: Completed | Type: Observational
Sponsor: InnFocus Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: INN005 - EXT
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Primary Open-angle Glaucoma
Keywords: POAG
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Trabeculectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- MicroShunt treatment group: Subjects previously randomized to this arm in pivotal study conducted under IDE G130028 were implanted with the device
  Interventions: Device: PRESERFLO® MicroShunt
- Trabeculectomy control arm: Subjects previously randomized to this arm in pivotal study conducted under IDE G130028 underwent trabeculectomy procedure
  Interventions: Procedure: Trabeculectomy

INTERVENTIONS:
Device: PRESERFLO® MicroShunt — Device surgically implanted
  Other Names: InnFocus MicroShunt® Glaucoma Drainage System
  Groups: MicroShunt treatment group
Procedure: Trabeculectomy — The procedure involves removal of a small portion of the trabecular meshwork and adjacent scleral tissue. Aqueous humor then drains into the subconjunctival space, creating a bleb on the external part of the eye, where it diffuses away.
  Groups: Trabeculectomy control arm

SUMMARY:
This prospective, concurrent controlled, open-label, multicenter study is designed to collect additional safety data through 5 years of follow-up for subjects randomized to either the treatment arm (PRESERFLO® MicroShunt with MMC) or the control arm (Trabeculectomy with MMC) of the INN-005 clinical study.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the long-term safety of the PRESERFLO® MicroShunt in subjects with Primary Open-Angle Glaucoma who have completed their Month 24 Follow-Up Visit in the INN-005 clinical study, by collecting safety data through 5 years post-operative follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has completed their Month 24 Follow-Up Visit in the INN-005 clinical study conducted under IDE G130028.
2. Subject was randomized into the INN-005 study and received the PRESERFLO® MicroShunt device or trabeculectomy. (Subjects who have had the device explanted, or replaced with another device, may be included).
3. Subject is willing and able to comply with all study requirements, including signing an informed consent form.

Exclusion Criteria:

1. Subject has exceeded the timeframe for the Month 60 Follow-Up Visit prior to enrollment for participation in this long-term follow-up study.

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes all living subjects who have completed the Month 24 Follow-Up Visit of the INN-005 clinical study after randomization to either the PRESERFLO® MicroShunt treatment arm or the Trabeculectomy control arm, and who are willing and able to extend their study participation and return for up to three (3) additional annual follow-up visits through post-operative Month 60. Up to 629 subjects may be enrolled at up to 24 sites located in the United States and at up to 5 sites located in Europe
Sampling Method: Non-Probability Sample
Enrollment: 279 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Palmberg, MD, PhD, Study Director — Bascolm Palmer Eye Institute
Locations (23):
- United States (19):
  - Arizona Advance Eye Research Institute, LLC., Glendale, Arizona
  - Vold Vision, Fayetteville, Arkansas
  - UCLA Medical Center Jules Stein Eye Institute, Los Angeles, California
  - University of California at Davis Eye Center, Sacramento, California
  - Ophthalmic Consultants of Connecticut, Meriden, Connecticut
  - Intermountain Eye Center, Eagle, Idaho
  - Eugene and Marilyn Glick Eye Institute, Indianapolis, Indiana
  - Stiles Eye Care Excellence & Glaucoma Institute, Overland Park, Kansas
  - Minnesota Eye Consultants, PA, Bloomington, Minnesota
  - New York Eye and Ear Infirmary of Mt. Sinai, New York, New York
  - Glaucoma Consultants of the Capital Region, Slingerlands, New York
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Ophthalmic Surgeons and Consultants of Ohio, Columbus, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Ophthalmic Partners of Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Glaucoma Associates of Texas, Dallas, Texas
  - Ophthalmology Associates, Fort Worth, Texas
  - University Eye Associates, Houston, Texas
  - R&R Eye Research, LLC, San Antonio, Texas
- Pôle Ophtalmologique de la Clinique Mutualiste, Pessac, Bordeaux, France
- A. O.U.P (Azienda Ospedaliere Universitaria Pisana) Stabilimento di Cisanello, Pisa, Cisanello, Italy
- Hospital Clínico San Carlos, Madrid, Spain
- Moorfields Eye Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This report presents data for 279 of subjects that completed the INN-005 Month 24 visit in the Phase II Pivotal Study who were enrolled in the INN-005 EXT study.
Groups:
- MicroShunt Treatment Group: Subjects previously randomized to this arm in pivotal study conducted under IDE G130028 were implanted with the device PRESERFLO® MicroShunt: Device surgically implanted
- Trabeculectomy Control Arm: Subjects previously randomized to this arm in pivotal study conducted under IDE G130028 underwent trabeculectomy procedure Trabeculectomy: The procedure involves removal of a small portion of the trabecular meshwork and adjacent scleral tissue. Aqueous humor then drains into the subconjunctival space, creating a bleb on the external part of the eye, where it diffuses away.
Period: Overall Study
Arm/Group | MicroShunt Treatment Group | Trabeculectomy Control Arm
Started | 217 | 62
Completed | 198 | 58
Not Completed | 19 | 4
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Death | 3 | 0
Not completed — Lost to Follow-up | 6 | 1
Not completed — 2 PRESERFLO Early Exit 1 PRESERFLO PI decision 1 PRESERFLO Study Exit | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MicroShunt Treatment Group | Trabeculectomy Control Arm | Total
Number analyzed (Participants) | 217 | 62 | 279
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 103 | 25 | 128
  >=65 years | 114 | 37 | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 27 | 138
  Male | 106 | 35 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 8 | 24
  Not Hispanic or Latino | 201 | 54 | 255
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 43 | 6 | 49
  White | 169 | 52 | 221
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 174 | 51 | 225
  Italy | 5 | 1 | 6
  United Kingdom | 4 | 2 | 6
  France | 11 | 1 | 12
  Spain | 11 | 2 | 13
  Netherlands | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Sight-threatening Adverse Events
Description: Sight-threatening Adverse events (AEs) that were started after enrollment in the INN-005-EXT study through Month 60.
Time Frame: Month 36 thru Month 60
Population: Incidence of sight-threatening adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | MicroShunt Treatment Group | Trabeculectomy Control Arm
Number analyzed (Participants) | 217 | 62
Participants | 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious Adverse Events (SAEs) were reported for all events that started after enrollment in the INN-005 EXT study through Month 60.
Description: Any untoward medical occurrence, unintended disease orinjury or any untoward clinical signs (including an abnormallaboratory finding) in subjects, users or other personswhether or not related to the investigational medical device.
Arm/Group | MicroShunt Treatment Group | Trabeculectomy Control Arm
All-Cause Mortality (participants affected / at risk) | 3/217 | 0/62
Serious Adverse Events (participants affected / at risk) | 8/217 | 0/62
Other Adverse Events (participants affected / at risk) | 172/217 | 47/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MicroShunt Treatment Group (N=217) | Trabeculectomy Control Arm (N=62)
Choroidal Hemorrhage (Eye disorders) | 1 (1) | 0 (0)
Erosion of the Device through the Conjunctiva (Eye disorders) | 4 (4) | 0 (0)
Central Retinal Artery Occlusion (Eye disorders) | 1 (1) | 0 (0)
Pseudophakic Bullous Keratopathy (Eye disorders) | 1 (1) | 0 (0)
Endothelial Cell Loss (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MicroShunt Treatment Group (N=217) | Trabeculectomy Control Arm (N=62)
Worsening in the Visual Field Mean Deviation (Eye disorders) | 54 (54) | 11 (11) — Confirmed Worsening in the Visual Field Mean Deviation (MD) ≥2.5dB compared to MD
Increased IOP Requiring Treatment (Eye disorders) | 57 (57) | 5 (5)
Cataract Progression (Eye disorders) | 35 (35) | 12 (12)
Loss 2 or More Lines of BCVA (Eye disorders) | 20 (20) | 4 (4) — Loss 2 or More Lines of BCVA on 2 Consecutive Standard Follow-ups 90 Days or more after Implantation (excluding Posterior Capsule Opacification, followed by post Nd: YAG Capsulotomy and improvement)
Posterior Capsule Opacification (Eye disorders) | 11 (11) | 6 (6)
Ptosis (Eye disorders) | 8 (8) | 7 (7)
Bleb Related Complications (Eye disorders) | 11 (11) | 3 (3) — Bleb Related Complications e.g. cystic bleb, flat bleb
Encapsulated Bleb (Eye disorders) | 10 (10) | 4 (4)
Hypotony (Eye disorders) | 6 (6) | 8 (8) — Hypotony (IOP <6mmHg at any Time)
Diplopia (Eye disorders) | 11 (11) | 1 (1)
Dry Eye (Eye disorders) | 28 (28) | 14 (14)
Epiretinal Membrane (Eye disorders) | 4 (4) | 5 (5)
Meibomian Gland Disease (Eye disorders) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT04333433/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT04333433/SAP_001.pdf